CLINICAL TRIAL: NCT07289386
Title: Effect of Instrument-assisted Soft Tissue Mobilization on Gait in Children With Spastic Diplegia
Brief Title: Effect of IASTM in Children With Diplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Elsayed Abbass, Assistant Proffessor of Pediatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005090
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral palsy; Gait
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): which received IASTM therapy in addition to the selected physical therapy program
  Interventions: Procedure: IASTM therapy in addition to the selected physical therapy program
- Control group (Active Comparator): which received selected physical therapy program
  Interventions: Procedure: selected physical therapy program

INTERVENTIONS:
Procedure: IASTM therapy in addition to the selected physical therapy program — The designed IASTM therapy was applied for 8-10 minutes per session, three times per week (every other day), for six successive weeks in addition to the selected physical therapy program was applied for one hour per session, three times per week (every other day), for six successive weeks
  Arms: Study group
Procedure: selected physical therapy program — The selected physical therapy program was applied for one hour per session, three times per week (every other day), for six successive weeks
  Arms: Control group

SUMMARY:
The aim was to evaluate the effect of using IASTM on passive ROM of the lower limbs and joint angles during gait in children with spastic diplegic CP. Methods: Thirty children with diplegic CP were randomly divided into 2 groups: a control group (which received a selected physical therapy program) and the study group (which received IASTM therapy in addition to the selected physical therapy program). They were treated three times weekly for six weeks. Passive ROM and active ROM during gait were assessed using a digital goniometer and Kinovea analysis software, respectively, before and after the proposed treatment period.

DETAILED DESCRIPTION:
Methods: Thirty children with diplegic CP were randomly divided into 2 groups: a control group (which received a selected physical therapy program) and the study group (which received IASTM therapy in addition to the selected physical therapy program). They were treated three times weekly for six weeks. Passive ROM and active ROM during gait were assessed using a digital goniometer and Kinovea analysis software, respectively, before and after the proposed treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 5 to 8 years old.
* spasticity ranged from 1 to 1+, according to Modified Ashworth Scale
* Children at level II according to Gross Motor Function Classification System
* They achieved independent walking with or without assistive device
* able to follow instructions and understand commands.

Exclusion criteria:

* Fixed muscle contractures or fixed bone deformities in the lower limb.
* Botox injection for the last six months.
* Orthopedic surgeries for the last year.
* Children with infectious diseases.
* Skin infection, seizures, and any lower limb soft tissue injury.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Active range of motion | six weeks
  measured by 2D gait analysis

SECONDARY OUTCOMES:
passive range of motion | six weeks
  measured by a digital goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Mai E. Abbass, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No